CLINICAL TRIAL: NCT02739165
Title: Phase III Clinical Study of ART-123 for the Treatment of Acute Exacerbation of Idiopathic Pulmonary Fibrosis: a Multicenter Randomized Placebo-controlled Double-blind Study to Assess the Efficacy and Safety of ART-123
Brief Title: Clinical Study of ART-123 for the Treatment of Acute Exacerbation of Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asahi Kasei Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ART-123-AEIPF-301
Record Dates: First submitted 2016-04-01; First posted 2016-04-15 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2017-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Acute exacerbations; Idiopathic pulmonary fibrosis; Recombinant human soluble thrombomodulin; ART-123
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — ART123

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- ART-123 (Experimental)
  Interventions: Drug: ART-123
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ART-123 — 380 U/kg/day by intravenous drip infusion in addition to standard of care steroid therapy
  Arms: ART-123
Drug: Placebo — Placebo by intravenous drip infusion in addition to standard of care steroid therapy
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of the intravenous drip infusion of ART-123 in patients with acute exacerbation of idiopathic pulmonary fibrosis (IPF) in a multicenter, double-blind, randomized, placebo-controlled, parallel group comparison study, and to confirm its superiority over placebo with survival rate on Day 90 as the primary endpoint.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients diagnosed with IPF who meet all criteria from (1) through (4) during the course of IPF
* (1)Unexplained development or worsening of dyspnea within 1 month during the course of IPF
* (2)Finding of new, bilateral ground glass opacities and/or consolidation on HRCT
* (3)No apparent Pulmonary infections, pneumothorax, malignant tumors, pulmonary embolism, or left heart failure
* (4)A decrease* in PaO2 of ≥10 mmHg or SpO2 of ≥4% under the same conditions compared with the level at the previous measurements

  * (*) In cases where no PaO2 or SpO2 test values under the same conditions are available, a patient with a P/F ratio ≤300 in the current episode of acute exacerbation is considered to have met criterion (4)
* Aged 40 years or older and no older than 85 years at the time of informed consent with either sex

Main Exclusion Criteria:

* Have intracranial hemorrhage, pulmonary hemorrhage, gastrointestinal bleeding (continued hematemesis, bloody discharge, gastrointestinal ulcer-induced hemorrhage)
* Have a history of cerebrovascular disorder (e.g., cerebral hemorrhage or cerebral infarction) within 52 weeks (364 days) before informed consent
* Patients for whom the completion of hemostatic treatment has not been confirmed after undergoing surgery of the central nervous system or after trauma
* Have a high risk for fatal or life-threatening hemorrhage
* Patients with malignant tumors
* Have acute exacerbation attributable to drug induced pulmonary disorder, after surgery for malignant tumors, chemotherapy, or radiation therapy
* Have acute exacerbation due to a thoracic surgical procedure (including thoracoscopic lung biopsy)
* Have a history of acute exacerbation of IPF
* Receiving mechanical ventilation through intratracheal intubation
* Patients who are pregnant or nursing, or who may be pregnant
* Patients with a platelet count less than 100,000/uL at the time of enrollment
* Patients with severe renal (serum Cr: ≥4 mg/dL) or hepatic (AST/ALT: ≥500 IU/L or T-Bil: ≥10 mg/dL) dysfunction
* Have been administered a commercially available thrombomodulin alfa (recombinant )(Recomodulin® for Intravenous Injection 12800) within 30 days before the start of investigational product administration
* Have a history of hypersensitivity for investigational product

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-05; Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Survival rate on Day 90 | 90 days

SECONDARY OUTCOMES:
Overall survival | 180 days after the start of investigational product administration in the last subject
Survival time up to Day 90 | 90days
P/F ratio | 4 days, 7 days, 15 days, 28 days, 60 days, 90 days
Coagulation tests | 4 days, 7 days, 15days, 28 days, 60 days, 90 days

OTHER OUTCOMES:
Chest imaging findings (chest HRCT findings) | Within 90days
Blood gas test | Within 90days
mMRC | Within 90days
CAT | Within 90days
Dyspnea-12 | Within 90days
Duration of respiration management | Within 90days
Inflammatory markers | Within 90days
Interstitial pneumonia markers | Within 90days
Total duration of respiratory system-related inpatient hospitalization | Within 90days
Adverse events (AEs) | Within 90days
AEs related to hemorrhage | Within 90days
Routine laboratory tests | Within 90days
Vital signs | Within 90days
Presence of anti-drug antibodies | Within 90days

CONTACTS AND LOCATIONS:
Overall Officials: Asahi Kasei Pharma Corporation, Study Chair — Asahi Kasei Pharma Corporation
Locations (26):
- Japan (26):
  - Nagoya, Aichi-ken
  - Seto, Aichi-ken
  - Kamogawa, Chiba
  - Sakura, Chiba
  - Kurume, Fukuoka
  - Ōgaki, Gifu
  - Himeji, Hyōgo
  - Kobe, Hyōgo
  - Naka, Ibaragi
  - Yokohama, Kanagawa
  - Sendai, Miyagi
  - Tenri, Nara
  - Kurashiki, Okanaya
  - Sakai, Osaka
  - Sayama, Osaka
  - Hamamatsu, Shizuoka
  - Shimotsuke, Tochigi
  - Bunkyo, Tokyo
  - Minato, Tokyo
  - Ōta-ku, Tokyo
  - Shibuya City, Tokyo
  - Shinjuku, Tokyo
  - Chiba
  - Fukuoka
  - Kumamoto
  - Nagasaki

REFERENCES:
- [Derived] Kondoh Y, Azuma A, Inoue Y, Ogura T, Sakamoto S, Tsushima K, Johkoh T, Fujimoto K, Ichikado K, Matsuzawa Y, Saito T, Kishi K, Tomii K, Sakamoto N, Aoshima M, Araya J, Izumi S, Arita M, Abe M, Yamauchi H, Shindoh J, Suda T, Okamoto M, Ebina M, Yamada Y, Tohda Y, Kawamura T, Taguchi Y, Ishii H, Hashimoto N, Abe S, Taniguchi H, Tagawa J, Bessho K, Yamamori N, Homma S. Thrombomodulin Alfa for Acute Exacerbation of Idiopathic Pulmonary Fibrosis. A Randomized, Double-Blind Placebo-controlled Trial. Am J Respir Crit Care Med. 2020 May 1;201(9):1110-1119. doi: 10.1164/rccm.201909-1818OC. PMID 31917621